CLINICAL TRIAL: NCT05246852
Title: The Effect of Training Provided According to the Health Promotion Model on Healthy Lifestyles and Self-efficacy in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hakan Avan (Other)
Responsible Party: Sponsor-Investigator, Hakan Avan, Instructor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: "hakanavan-0001
Record Dates: First submitted 2022-01-29; First posted 2022-02-18 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Adolescent Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: healthy lifestyle education
- control group (No Intervention)

INTERVENTIONS:
Behavioral: healthy lifestyle education — A total of 6 sessions on physical activity, nutrition, substance abuse, sexual life, check-up, accidents and injuries will be organized for the adolescents in the intervention group. The sessions will be organized every other week. Each session will be conducted in three stages. First Stage: The researcher will provide training on the subject of the session for nearly 15 minutes. Second Stage: The researcher will show animation film (nearly 3 to 5 minutes) developed by him/her related to the session. Third Stage: Groups of six will be created for the Philips 66 technique application and a spokesman will be chosen. Each group will have an online meeting and discuss the session subject in six minutes under the administration of the researcher. The spokesman of each group will present the discussion outcome in the big group meeting at the end of the discussion. The researcher will summarize the subject after the presentation of each spokesman and terminate the session.
  Arms: intervention group

SUMMARY:
The study was designed as a randomized controlled experimental study in a pretest-posttest design to determine the effect of training provided according to the health promotion model concerning the factors which affect healthy lifestyle in adolescents, on health promotion behavior. It is aimed for adolescents to take health responsibility by increasing their self-efficacy levels and make it a part of their lives. The sample will consist of 72 adolescents (36 in intervention group, 36 in control group) at significance level of 5%, power of 80% and effect size of 0.5-0.75 in a population including 45.737 adolescents aged 14 to 17 years in schools affiliated with Kahramanmaraş Provincial Directorate for National Education. In the first stage of determining the sample, two schools will be determined by drawing lots among the schools affiliated to the Provincial Directorate of National Education and the researcher will assign adolescents, who meet the inclusion criteria, to intervention (n=36) and control (n=36) groups from the first and second schools, respectively using the stratified sampling method and the random numbers table. The inclusion criteria will be being aged 14 to 17 years, speaking Turkish, having parental permission, having no mental or neurological disability and having no chronic illness. In the study, the randomization will be conducted according to age, gender, body mass index, department, and family type. The Adolescent and Parent Information Form (Socio-demographic Characteristics), the Adolescent Lifestyle Profile (ALP) and the Self-efficacy Scale (SES) will be used to gather the data. The data will be collected online from 72 adolescents receiving education in the two high schools affiliated with the Provincial Directorate for National Education between 14 February 2022 and 15 May 2022. The first measurements and trainings will be conducted online. In the first measurement, there will primarily be a meeting activity and then the data collection forms (Socio-demographic Characteristics, the ALS, the SES) will be collected online from the intervention and the control group via e-mail or social media applications. Following the first measurement, the first session will be conducted in the intervention group. As of the first session, a total of six sessions, one in every week will be conducted. In the final session where the applications finish, the posttest-1 including the data collection forms (Socio-demographic Characteristics, the ALS, the SES) will be used in the intervention and control groups. The posttest-2 including the same forms will be applied to the groups one month later. A preliminary application will be performed online in 10 adolescents who remain outside the sample and meet the inclusion criteria. According to the results obtained from the preliminary application, necessary arrangements will be made on the forms and the session and the application will be finalized. A total of 6 sessions on physical activity, nutrition, substance abuse, sexual life, check-up, accidents and injuries will be organized for the adolescents in the intervention group. The sessions will be organized every other week. Each session will be conducted in three stages. First Stage: The researcher will provide training on the subject of the session for nearly 15 minutes. Second Stage: The researcher will show animation film (nearly 3 to 5 minutes) developed by him/her related to the session. Third Stage: Groups of six will be created for the Philips 66 technique application and a spokesman will be chosen. Each group will have an online meeting and discuss the session subject in six minutes under the administration of the researcher. The spokesman of each group will present the discussion outcome in the big group meeting at the end of the discussion. The researcher will summarize the subject after the presentation of each spokesman and terminate the session. The nursing intervention according to the SGM will not be performed in the control groups. However, the adolescents will continue their routine training.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be being aged 14 to 17 years,
* speaking Turkish,
* having parental permission,
* having no mental or neurological disability,
* having no chronic illness.

Exclusion Criteria:

* Those who fill in the forms incompletely or incorrectly
* Those who do not want to participate in the research during the implementation phase of the research.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
develop their self-efficacy related to physical activity | through study completion, an average of 5 week
  Adolescent Lifestyle Profile and the Self-efficacy Scale
develop their self-efficacy related to healthy diet | through study completion, an average of 5 week
  Adolescent Lifestyle Profile and the Self-efficacy Scale
develop their self-efficacy related to protection from substance abuse | through study completion, an average of 5 week
  Adolescent Lifestyle Profile and the Self-efficacy Scale
develop their self-efficacy related to sexuality | through study completion, an average of 5 week
  Adolescent Lifestyle Profile and the Self-efficacy Scale
develop their self-efficacy related to check-up | through study completion, an average of 5 week
  Adolescent Lifestyle Profile and the Self-efficacy Scale
develop their self-efficacy related to accidents and injuries | through study completion, an average of 5 week
  Adolescent Lifestyle Profile and the Self-efficacy Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hakan Avan, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No